CLINICAL TRIAL: NCT02543905
Title: The PROFILE Study: Germline Genetic Profiling: Correlation With Targeted Prostate Cancer Screening and Treatment
Acronym: PROFILE
Status: Recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); University of Cambridge (Other); University of Oxford (Other); Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4045
Record Dates: First submitted 2015-07-13; First posted 2015-09-07 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Prostate Biopsy; Genetic Counselling; Genetic Markers
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, urine, DNA, RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family History Cohort: Men of any ethnicity with a family history of prostate cancer defined as:
  * Men with a first degree relative (or second degree if through female line) with histologically or death certificate proven PrCa diagnosed at <70 years
  * Men with two relatives on the same side of the family with histologically or death certificate proven PrCa where at least one is diagnosed at <70 years
  * Men with three relatives on the same side of the family with histologically or death certificate proven PrCa diagnosed at any age
  Interventions: Procedure: Prostate MRI and Biopsy
- Black African / Black African-Caribbean Cohort: Men of black African or black African-Caribbean ancestry defined as:
  Both parents and all 4 grandparents being of black African or black African-Caribbean ancestry.
  Interventions: Procedure: Prostate MRI and Biopsy
- High-risk gene mutation cohort: Men of any ethnicity with a genetic predisposition to having prostate cancer e.g., being known to have inherited a gene mutation that increases risk of prostate cancer (gene mutation including BRCA1, BRCA2, ATM, PALB2, MLH1, MSH2, MSH6, CHEK2 and other DNA repair gene mutations as listed in the study protocol); and/or being known to have a high polygenic risk score (PRS) (defined as being in the top tenth percentile prior to enrolment).
  Interventions: Procedure: Prostate MRI and Biopsy

INTERVENTIONS:
Procedure: Prostate MRI and Biopsy — All men will be offered a MRI and prostate biopsy and they can either opt to undergo these procedures at baseline irrespective of PSA level at baseline or they can undergo PSA-only screening until clinically indicated based on an age-defined PSA threshold, at which point, they will undergo prostate MRI and biopsy once their PSA reaches the threshold.

SUMMARY:
Prostate cancer is now the most common cancer in men in the Western world. In the United Kingdom (UK), there were over 52,000 new cases diagnosed in 2016-2018 and a lifetime risk of 1 in 8. Prostate cancer (PrCa) can run in some families and research studies have identified several genetic changes in Caucasian populations that are thought to increase the risk of developing prostate cancer. Other studies have shown that men from certain ethnic groups also have a higher risk of prostate cancer, and this includes men of black African or black African-Caribbean ancestry. This study aims to look at men with a higher risk of prostate cancer based on their ethnicity, family history and/or genetic predisposition to see whether any of these genetic changes are present in their DNA (genetic material) and whether this could be a helpful screening tool in prostate cancer screening programmes. It is thought that many genetic changes are involved in the development of prostate cancer and research is being carried out worldwide to identify these genetic changes. Some of these changes may cause a very slight increase in prostate cancer risk while others may cause a much larger increase in risk of developing prostate cancer. The investigators will invite (i) men of any ethnicity with a family history of prostate cancer; (ii) men of black African or black African-Caribbean ancestry; and (iii) men of any ethnicity with a known genetic predisposition to having prostate cancer (e.g., being known to have inherited a gene mutation that increases risk of prostate and/or being known to be in the top tenth percentile of the polygenic risk score (high PRS score prior to enrolment) for targeted prostate screening (Prostate Specific Antigen (PSA) testing, MRI and a biopsy of the prostate gland) and genetic profiling. The outcome of these prostate cancer screening investigations will be compared with the genetic profiles of those taking part in the study in order to look for certain genetic changes in the gene code that are thought to increase prostate cancer risk. This research will help us to determine what the role of such genetic profiling is in a prostate cancer screening programme and if it helps identify men at high prostate cancer risk.

DETAILED DESCRIPTION:
Purpose and Design

The aim of the PROFILE study is to investigate the role of targeted prostate cancer screening in men at a genetically higher risk to estimate the incidence of PrCa and the sensitivity and specificity of PSA screening in these populations and correlate this with genetic profiles and biological endpoints. Additionally, the study aims to identify biomarkers from biological samples (such as blood and urine) as well as imaging technologies (e.g. MRI and new imaging techniques) as predictive markers of the risk of developing PrCa and to correlate these with genetic risk. This study has been designed using an observational approach to look at the correlation of cancer incidence (on biopsy) with genetic profile. The aim is to evaluate targeted screening for prostate cancer in men at a genetically higher risk to estimate the incidence of prostate cancer and the sensitivity and specificity of PSA screening in these populations and correlate this with genetic profiles (i.e. single nucleotide polymorphism (SNP) profiles) and biological endpoints.

Three cohorts will be recruited:

1. Men of any ethnicity with family history of prostate cancer.
2. Men of black African or black African-Caribbean ancestry.
3. Men of any ethnicity with a genetic predisposition to having prostate cancer (e.g., being known to have inherited a gene mutation that increases risk of prostate cancer (i.e. high-risk gene mutation) and/or being known to have a high polygenic risk score (high PRS score) defined as being in the top tenth percentile prior to enrolment.

Men with no prior screening will be offered biopsy and genetic profiling. This will provide data on genetic profiling and correlation with biopsy irrespective of PSA in men who have not had any previous screening.

A PSA screening algorithm was considered as an alternative to biopsy but there is great controversy over the PSA threshold that should be used as a cut-off. Recent data have shown that a considerable percentage of men with a PSA within normal range have cancer at biopsy. Therefore, it was decided by the Steering Committee that all participants should be offered a biopsy within this study. This will tell us the acceptability of this approach.

Some men may opt not to have biopsy at baseline (i.e. initial stage). These men will be followed up with annual PSA, whereby prostate biopsy would be offered if PSA is above or equal to 1.0ng/ml if the man is aged under 50 years, or where PSA is above or equal to 2.0ng/ml if the man is aged fifty years or over.

Eligibility and Recruitment

Either:

(1) Men of any ethnicity with a positive family history of PrCa defined as:

* Men with a first degree relative (or second degree if through female line) with histologically or death certificate proven PrCa diagnosed at <70 years
* Men with two relatives on the same side of the family with histologically or death certificate proven PrCa where at least one is diagnosed at <70 years
* Men with three relatives on the same side of the family with histologically or death certificate proven PrCa diagnosed at any age

Or (2) Men of black African or black African-Caribbean ancestry defined as:

Both parents and all 4 grandparents being either black African or black African-Caribbean.

Or (3) Men of any ethnicity with a genetic predisposition to having prostate cancer e.g., being found to have inherited a gene mutation that increases risk of prostate cancer (e.g. BRCA1, BRCA2, ATM, PALB2, MLH1, MSH2, MSH6, CHEK2 and other DNA repair gene mutations as listed in the study protocol); and/or being known to have a high polygenic risk score (PRS) (defined as being in the top tenth percentile prior to enrolment).

* Age 40- 69 years
* WHO performance status 0-2
* Absence of any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow up schedule.

Exclusion criteria

* Previous cancer with a life expectancy of less than five years.
* Previous PrCa
* Negative biopsy within one year before recruitment
* Comorbidities making prostate biopsy risk unacceptable (anticoagulants or antiplatelet medication including Warfarin, Clopidogrel, Apixaban, Dabigatran or other NOAC (Novel Oral Anti-Coagulant); poorly controlled diabetes, cardiovascular/respiratory disease, immunosuppressive medication or splenectomy).
* Men with body mass index (BMI) 40 and above.
* Men with BMI 35 and above plus other co-morbidities.
* Contraindications to having an MRI (non-MRI compliant pacemakers, aneurysm clips, metallic cardiac valve/stent, Ventriculo-Peritoneal (VP) shunt, cochlear implant, neurotransmitter, metallic foreign bodies in eye(s), other metalwork, claustrophobia)
* Any significant psychological conditions that may be worsened or exacerbated by participation in the study

Subject Withdrawal

o Subjects may withdraw from the study at any time if they so wish without giving a reason. No further data will be collected about that individual, and any unused samples will be destroyed. Data collected up to that point will be retained for audit purposes.

Cancer cases Men who are found to have prostate cancer at biopsy will be referred to their local urologist for treatment according to local policy. Men will be followed up for 10 years in order to evaluate the different treatment regimens.

Genetic Profiling All men will have genetic profiling to correlate with disease status and men will be given the results of this test. It will be emphasised that these are research results and written information will be provided as a reference guide.

Informed Consent All subjects will be informed of the aims of the study, the possible adverse events, the procedures and possible hazards to which he will be exposed, and the mechanism of treatment allocation if prostate cancer was to be diagnosed. He will be informed as to the strict confidentiality of his patient data, but that his medical records may be reviewed for trial purposes by authorised individuals other than their treating physician.

It will be emphasised that participation in this study is voluntary and that the subject is allowed to refuse further participation in the protocol whenever he wants. This will not prejudice the subject's subsequent care. Documented informed consent will be obtained, according to the principals of good clinical practice (GCP), for all subjects included in the study before they are registered onto the study.

Risks, burdens, benefits There is a risk of complications from having a prostate biopsy, and these complications are detailed in the patient information sheet, together with likelihood of incidence. Complications are rare and standard procedures will be followed at all sites to minimise their occurrence. The benefit of taking part may be that prostate cancer may be diagnosed in men previously unaware that they had the disease. While there is the potential for overdiagnosis of indolent disease, there is also the potential for detecting and treating clinically significant disease.

Provision of results from the genetic profiling One further consideration is the occurrence of anxiety as a result of taking part in the study, particularly in receiving research genetic test results. There is considerable uncertainty about how genetic profile relates to predicted risk of prostate cancer. For this reason individualised written information will be provided to each participant putting the research results in the context of the current population risks. It will be stressed that these are research results only and that the investigators do not fully understand the meaning of the results.

A psychosocial study is being run concurrently and will explore these issues in more depth and the participant's experience of receiving these results will be an important component of the evaluation of this study.

Confidentiality All information which is collected will be accessible only to the immediate study team. Any data that is shared will be de-identified and any published data will be anonymised so that no participant is recognisable from the results.

Medical records and the data collected for the study may be looked at by authorised persons from the Institute of Cancer Research, by regulatory authorities and by authorised people to check that the study is being carried out correctly. All will have a duty of confidentiality to participants.

End of Study Follow-up After the participant has completed the study they will be advised about any ongoing screening or follow-up that is required. This will be organised through the participants general practitioner (GP).

Use of samples in future research The informed consent process will explain that samples are donated as a "gift". If any of the samples collected are to be considered for use in future research projects this would have to be approved by the Ethics Committee first.

ELIGIBILITY:
Inclusion Criteria:

Either:

1. Men of any ethnicity with a positive family history of PrCa defined as:

   * Men with a first degree relative (or second degree if through female line) with histologically or death certificate proven PrCa diagnosed at <70 years
   * Men with two relatives on the same side of the family with histologically or death certificate proven PrCa where at least one is diagnosed at <70 years
   * Men with three relatives on the same side of the family with histologically or death certificate proven PrCa diagnosed at any age

   Or
2. Men of black African or black African-Caribbean ancestry defined as:

   Both parents and all 4 grandparents being of either black African or black African-Caribbean ancestry.

   Or
3. Men of any ethnicity with a genetic predisposition to having prostate cancer e.g., being known to have inherited a gene mutation that increases risk of prostate cancer (e.g. BRCA1, BRCA2, ATM, PALB2, MLH1, MSH2, MSH6, CHEK2 and other DNA repair gene mutations as listed in the study protocol); and/or being known to have a high polygenic risk score (PRS) (defined as being in the top tenth percentile prior to enrolment).

   * Age 40- 69 years
   * WHO performance status 0-2
   * Absence of any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow up schedule.

Exclusion Criteria:

* Previous cancer with a life expectancy of less than five years.
* Previous PrCa
* Negative biopsy within one year before recruitment
* Co-morbidities making prostate biopsy risk unacceptable (anticoagulants or antiplatelet medication including Warfarin, Clopidogrel, Apixaban, Dabigatran or other NOAC (Novel Oral Anti-Coagulant); poorly controlled diabetes, cardiovascular/respiratory disease, immunosuppressive medication or splenectomy)
* Men with body mass index (BMI) 40 and above.
* Men with BMI 35 and above plus other co-morbidities.
* Contraindications to having an MRI (non-MRI compliant pacemakers, aneurysm clips, metallic cardiac valve/stent, Ventriculo-Peritoneal (VP) shunt, cochlear implant, neurotransmitter, metallic foreign bodies in eye(s), other metalwork, claustrophobia)
* Any significant psychological conditions that may be worsened or exacerbated by participation in the study

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 350 men in each cohort*
  *The family history cohort will overrecruit to a total of 800, until 350 participants undergo MRI & biopsy; both the Black and high-risk gene cohorts will overrecruit to a total of 400 participants each, to replace any participants who withdrew and/or any protocol non-compliant cases (e.g. those who underwent MRI but did not complete the biopsy).
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2015-03-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The association of specific genetic profiles and biomarkers to predict outcome of prostate screening in men at higher genetic risk | 5 years
  To investigate the role of targeted prostate cancer screening in men at higher genetic risk (i.e. family history, ethnicity, gene mutation status), its association with specific genetic profiles and biomarkers as predictive tools of the risk of developing prostate cancer and to correlate these with genetic risk.

SECONDARY OUTCOMES:
The incidence and aggressiveness of prostate cancer in men at higher genetic risk. | 5 years
  To determine the incidence and aggressiveness of prostate cancer in these men at a higher genetic risk.
The association of Diffusion Weighted MRI (DW-MRI) findings with prostate biopsy results. | 5 years
  To determine whether imaging techniques such MRI can be used to identify prostate cancer when compared to prostate biopsy results.
The incidence of abnormal imaging (using 3D ultrasound combined with shear wave elastography) and correlation with biopsy outcome and to correlate standard 12 core prostate biopsies with targeted biopsies based on abnormalities identified at DWMRI. | 5 years
  To determine the incidence of abnormal imaging at MRI in correlation with biopsy outcome.
The association of biological sample biomarker profiles with prostate biopsy result. | 5 years
  To identify biomarkers from biological samples and determine their association with prostate biopsy result.
The association of quantitative imaging biomarkers with prostate biopsy result | 5 years
  To identify imaging biomarkers and determine their association with prostate biopsy result.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind A Eeles, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- Institute of Cancer Research and Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be applied for via the Data Access Committee

REFERENCES:
- See also: Cancer Research UK (2022) — https://www.cancerresearchuk.org/health-professional/cancer-statistics-for-the-uk